CLINICAL TRIAL: NCT05156645
Title: An Adaptive Phase I/II/III Trial to Evaluate the Efficacy and Safety of Anti-SARS-CoV-2 Monoclonal Antibody Combination (SCTA01C and SCTA01) for Treatment of Outpatients With COVID-19
Brief Title: A Study to Evaluate Efficacy and Safety of the Combination of SCTA01 & SCTA01C in Outpatients With COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was withdraw due to the fast spread of Omicron variant worldwide
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCTA01/SCTA01C-A301
Record Dates: First submitted 2021-12-09; First posted 2021-12-14 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — upanovimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCTA01 and SCTA01C+SOC (Experimental)
  Interventions: Drug: SCTA01 and SCTA01C
- Placebo+SOC (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCTA01 and SCTA01C — Diluted by 0.9% normal saline
  Arms: SCTA01 and SCTA01C+SOC
Drug: Placebo — Diluted by 0.9% normal saline
  Arms: Placebo+SOC

SUMMARY:
The study is comprised of two parts: safety evaluation part (Phase I/II) and the pivotal study (Phase III) to evaluate the efficacy and safety of the combination of SCTA01 & SCTA01C compared to placebo in addition to Standard of Care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female adults, ≥18 years old of age at the time of randomization;
* Participants should have at least one of COVID-19 risk factor;
* Participants should have at least 2 COVID-19 related symptoms;
* Has symptoms consistent with COVID-19 as determined by the investigator with onset ≤10 days before randomization;
* First positive SARS-CoV-2 viral infection tested (PCR or antigen-based diagnostic tests) in samples collected ≤5 days prior to start of the infusion;

Exclusion Criteria:

* Participants with a history of severe anaphylaxis, such as severe anaphylactic reaction, urticaria, and angioedema;
* Have SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300, respiratory rate ≥30 per minute, heart rate ≥125 per minute (FDA);
* Require mechanical ventilation or anticipated impending need for mechanical ventilation;
* Suspected or proven serious bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking part in this study;
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experience COVID-19 related hospitalization (defined as at least 24 hours of acute care) or death (all cause) up to Day 29 (Phase III) | Day 29
Proportion of patients with ≥Grade 3 treatment related adverse event (TRAE) up to Day 8 (Phase I/II) | Day 8

SECONDARY OUTCOMES:
Time to sustained resolution of all COVID-19-related symptoms | Day 29
Change in symptom score (total of ratings) | Day 3, 5, 7, 11, 15, 22, and 29
Time to symptom improvement | Day 29
Proportion of participants that achieve SARS-CoV-2 clearance in NP or OP samples | Day 29
Immunogenicity assessment includes the number and percentage of patients who develop detectable anti drug antibody | Day 120
Mean concentration-time profiles of SCTA01 and SCTA01C | Day 120

IPD SHARING:
Plan to Share IPD: Yes